CLINICAL TRIAL: NCT02754258
Title: The Effects of Methylphenidate on the Reduction of Food Energy Intake and on the Augmentation of Energy Expenditure
Brief Title: The Effects of Methylphenidate on Energy Intake and Energy Expenditure
Acronym: MPH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: University of Ottawa (Other)
Responsible Party: Principal Investigator, Phillippe Robaey, Qualified Investigator, MD, PhD, FRCPC, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15/10E
Record Dates: First submitted 2016-04-12; First posted 2016-04-28 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — 5,10-dihydro-5-methylphenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 60 day oral administration of sugar placebo twice per day before lunch and supper.
  Interventions: Drug: Placebo
- Methylphenidate (MPH) (Experimental): 60 day oral administration of active study drug (methylphenidate) twice per day before lunch and supper.
  Interventions: Drug: MPH

INTERVENTIONS:
Drug: MPH — 60 days on oral methylphenidate administered 2 times daily before lunch and supper.
  Other Names: pms-Methylphenidate
  Arms: Methylphenidate (MPH)
Drug: Placebo — 60 days on oral placebo administered 2 times daily before lunch and supper
  Other Names: Sugar Placebo
  Arms: Placebo

SUMMARY:
The Problem: Obesity is one of the leading causes of chronic disease and death. The efficacy of diet and exercise to sustain weight loss over the long term is weak. While pharmacotherapy is more effective than behavior intervention in maintaining weight loss the effects are often not sufficient to achieve optimal health benefits. Current drug treatments may be sub-optimal because they do not directly target the rewarding value of food, drive to eat, food liking, and impulsivity for eating energy dense snack foods, all of which influences both quantity and quality of food intake and impacts adherence needed to maintain weight loss.

The Solution: The limitations in current anti-obesity agents are potentially addressed by Methylphenidate (MPH). We showed that MPH reduces food intake, dietary fat intake, hunger and food reward, as increase resting energy expenditure in obese and non-obese adults;however, no controlled field trials have been conducted in obese individuals without ADHD.

Objectives/Hypotheses: Primary: To test the effects of MPH on energy intake in obese men and women. Secondary: to examine the effects of MPH on energy expenditure, body weight, impulsivity, food reward, and olfaction. The investigators predict that compared to placebo, MPH will show reduced appetite, along with reduced impulsivity, food reward, and smell function.

Deliverable: This study may be the first to establish the short-term efficacy and safety of using MPH for weight loss, and if successful, data will inform a larger trial that can potentially identify MPH as a novel therapeutic agent for treating obesity and related chronic diseases in a predisposed population.

DETAILED DESCRIPTION:
Research Objectives and Hypotheses

Primary: The primary objective of this study is to examine whether Methylphenidate (MPH) at dose of 0.50 mg/kg (not exceeding 100 mg/day) can lead to a sustained reduction in energy intake in obese adolescents and adults. Based on the investigators' pilot data in adults, it is predicted that daily administration of MPH for 60 consecutive days will produce reductions in food intake (both in lab and free-living) compared to placebo, extending our previous findings to a longer period of time and to obese adolescents. Prior to beginning the intervention, both MPH and placebo treatment groups will receive lifestyle advice (eating and exercise guidelines for healthy living). The primary outcome measures will rely on the validated measurements of energy intake (in lab lunch buffet and out of lab 3 day food menu).

Secondary objectives/hypotheses: The effects of MPH on all components of energy expenditure will be investigated. Based on the investigators' pilot data, it is predicted that from Baseline to 60 days, MPH will increase total energy expenditure (TEE) when compared with placebo, mostly through greater resting energy expenditure (REE) and thermic effects of food (TEF). It is hypothesized that after the 60-day intervention the MPH group will experience a significantly attenuated reduction in REE compared to placebo. We predict that the MPH group will lose body weight at 2 months, whereas, it is predicted that there will be no change in body weight for the placebo. The investigators will also explore the effects of MPH on macronutrient preference and consumption, and on the rewarding value of energy dense snack foods. Based on previous findings, the investigators predict that MPH will reduce consumption of energy dense, high fat/sugar foods but have little effect on consumption of foods low in calories, fats or sugars. In addition, it is predicted that the reduction in intake of energy dense, high fat/sugar foods will be mediated by reductions in the rewarding value of food and impulsivity as measured by well validated computerized simulations. Also explored will be the effects of MPH on olfaction and it is predicted that compared to placebo, individuals taking MPH will have reduced smell function. It is also predicted the MPH group will show reduced appetite sensations, reduced rewarding value of food, reduced impulsivity for snack food, and reduced palatability ratings of food compared to placebo at 2 months.

Trial Design

The trial design will consist of a randomized, double blind, placebo-controlled 2 parallel arm study. The two randomly assigned treatment groups will consist of administrating a placebo or short-acting MPH two-times daily 1 hour before meals for a period of 2 months (60 consecutive days). Prior to being randomized into either the placebo group or the experimental (MPH) group, subjects will first have had to respond to a recruitment poster, newspaper advertisement. Once it is determined with that initial screening that the participant still meets inclusion criteria, they will be invited to come to the laboratory for a screening visit to determine whether they meet eligibility criteria, to sign informed consent, and to take a test dose of MPH in order for a nurse to closely monitor any potential side-effects prior to starting the 2-times daily dosing of MPH or placebo.

Trial Procedures

The proposed study will consist of six visits to the laboratory for a total of twenty-four hours, as follows: there will be an initial clinical screening visit (4 hrs), three repeated measures test days (6hrs each; two at baseline and one at 60 days), a mid-point visit (1hr), and a Lunch Box visit (10 minutes to obtain out of laboratory food). School-aged participants will not have to miss school to participate; if necessary, testing will be able to be performed over the course of the weekend. After the initial laboratory visit and informed consent (i.e. clinical screening visit), participants will be randomized at the Baseline 1 visit to one of two treatment groups to either receive placebo or MPH two times daily for a 2 month intervention period that starts at the Baseline 2 visit. In order to track physical activity energy expenditure, participants will be instructed to wear accelerometers for 1 week between the in lab screening visit and the Baseline 1 visit, and then again while under MPH or placebo for 1 week between the mid-point visit and the Final repeated measures test day. Upon leaving the Baseline 1 test day (i.e. no drug or placebo) participants will receive a 3 day supply of food from which they will exclusively eat from until they return to the lab 4 days later for the Baseline 2 repeated measures test day (i.e. under drug or placebo). Similarly, 4 days prior to the Final repeated measures test day, participants will again have to visit the laboratory for their "Lunch Box" visit to obtain their three days' supply of food from which they will eat exclusively from. Participants will return to the laboratory to complete the study at the Final (day 60) repeated measures test day after 3 days of eating from the "Lunch Boxes". For the 1 hour mid-point visit (at day 30) participants will be weighed and will report any perceived side-effects from the MPH or placebo. At this mid-point visit participants will bring in their pill container to verify compliance and to receive final 30 day supply of drug or placebo. At this time participants will be asked if they have begun any new medication or have started any over-the-counter medication as part of the study's safety monitoring protocol. A side-effects check list will also be provided to the participants upon leaving the Baseline 2 testing session; participants will be informed to note any perceived side-effects nightly for the first 14 days being on the study medication and will be instructed to notify the study coordinator as soon as specific side-effects are noted as being Major.

Consent and Clinical Screening

Initial Screening Visit (4 hours)

Before beginning the study, a meeting between the study coordinator and the participant will occur in order to get consent and in order for the participant to ingest a test dose of MPH under the supervision of a nurse. The study coordinator will contact the participant in order to arrange a time for the approximately 4 hour meeting. The weight and height (thus BMI) will be measured upon arrival. The participant will then have to respond to questionnaires, e.g. the Wender-Utah Rating Scale (to assess traits compatible with ADHD), the Beck Depression Inventory (to assess depressive symptoms), the "Three-Factor Eating Questionnaire" (to assess eating style) and the Drug Abuse Screening Test (to ensure no underlying drug problem). If the participant is a female they cannot be pregnant to be included in the study; thus a pregnancy test will be administered and if it is determined that they are pregnant they will be referred to visit their family physician and excluded from the study. If eligible, the participant will be asked to read and sign the consent form. Eligible participants will then see a nurse who will administer the all of the measures outlined in the Case Report Form, e.g., a physical exam, medical history assessment, baseline vital signs, electrocardiogram (ECG), etc. The nurse will then administer a test dose of 0.5mg/kg of MPH and for a period of three hours after the ingestion of MPH the nurse will closely monitor any potential side-effects of the drug by measuring heart rate, blood pressure, and by following a detailed side-effects check-list. If at any point the participant rates and of the side effects as "Prohibitive", then he/she will be excluded from the study. The participant will also be excluded from entering the study if they demonstrate an abnormal ECG systolic or if blood pressure exceeds the baseline reading by 20mmHg or if diastolic blood pressure exceeds the baseline reading by 10mmHg, BP > 160/100, or resting pulse increased by 20 beats/minute from the baseline. As part of the comprehensive safety assessment to determine eligibility, the ECG data file that is collected will be stored via a USB external hard drive and then sent to CHEO cardiology to be read by a cardiologist. Once it is determined by the cardiologist that the ECG rhythm is normal, both the cardiologist and the QI will sign off on the Case Report form, indicating that the participant is eligible for enrollment. If it is determined by the ECG reading that the participant is not eligible, they will be called up by the study coordinator and told of the incidental findings and subsequently informed to visit their family physician to follow-up. The participant may bring the consent form home to further study its content before signing it. Prior to leaving the initial screening visit participants will be instructed on how to strap on an omni-directional accelerometer and instructed on how to fill out the log sheet which gathers information on when the monitors are worn and when they are taken off, which is needed to evaluate wear time for a seven day period. Participants will be instructed to return the accelerometers at their next visit, Baseline 1.

Free and informed Consent

During the initial screening visit, if a candidate meets the inclusion criteria, the coordinator will explain the research protocol to the subject. This will be done in order to explain in detail the requirements of the protocol and to answer all the questions from potential participants. If potential participants are still interested to participate in the study, the coordinator will then distribute, explain and answer questions regarding the consent form to the participant. The participant will then be asked to sign the informed consent letter.

Active Investigational Product Description

pms-METHYLPHENIDATE (methylphenidate hydrochloride) is a racemate consisting of a 1:1 mixture of d-methylphenidate (d-MPH) and l-methylphenidate (l-MPH). pms-METHYLPHENIDATE is a mild central nervous system stimulant with more prominent effects on mental than motor activities. The mode of action in man is not completely understood, but its stimulant effects are thought to be due to cortical stimulation and possibly to stimulation of the reticular activating system. There is neither specific evidence which clearly establishes the mechanism whereby methylphenidate produces its mental and behavioural effects in children, nor conclusive evidence regarding how these effects relate to the condition of the central nervous system (CNS). Methylphenidate hydrochloride is rapidly and extensively absorbed from the tablets following oral administration; however, owing to extensive first-pass metabolism, bioavailability is low (approx. 30%) and large individual differences exist (11-52%). Peak plasma concentrations of 10.8 and 7.8 ng/mL were observed, on average, 2 hours after administration of 0.30 mg/kg in children and adults, respectively. Methylphenidate is eliminated from the plasma with a mean half-life of 2.4 hours in children and 2.1 hours in adults. The apparent mean systemic clearance after an oral dose is 10.2 and 10.5 L/h/kg in children and adults, respectively for a 0.3 mg/kg dose, and 0.565 L/h/kg after an intravenous dose of the racemate in healthy adult volunteers. These data indicate that the pharmacokinetics of methylphenidate in hyperactive children is similar to that in healthy adult volunteers. The apparent distribution volume of methylphenidate in children was approximately 20 L/kg, with substantial variability (11-33 L/kg). The volume of distribution after an intravenous dose (Vss) is 2.23 L/kg for the racemate in healthy adult volunteers.

Following oral administration of methylphenidate, 78-97% of the dose is excreted in the urine and 1-3% in the feces in the form of metabolites within 48-96 hours. The main urinary metabolite is ritalinic acid (a-phenyl-2-piperidine acetic acid, PPAA); unchanged methylphenidate is excreted in the urine in small quantities (<1%). Peak PPAA plasma concentrations occurred at approximately the same time as peak methylphenidate concentrations, however, levels were several-fold greater than those of the unchanged drug. The half-life of PPAA was approximately twice that of methylphenidate.

Role of CHEO Pharmacy

Section C.05.010 of the Division 5 Regulations pertains to the sponsor's (i.e. Children's Hospital of Eastern Ontario) obligations in regards to Good Clinical Practice. The CHEO pharmacy will have the following obligations-compliant with said Regulations-with respect to the drug/placebo management: drug acquisition and dispensing, maintenance of inventory and accountability and reconciliation of records, labelling of study medication, storage of inventory, and general records such as patient information forms and creating patient binders. Note that in Division 5, Health Canada mandates that records must be maintained for a period of 25 years, and the CHEO pharmacy will ensure the maintenance of such record keeping.

Safety Assessments and Trial Monitoring

Clinical Safety Assessments

The following assessments will be performed to determine the safety of MPH Hydrochloride: vital signs (blood pressure and pulse); monitoring effects/symptoms (side effects checklist). Those who report or show heightened blood pressure or heart rate side effects from the test doss of MPH at the clinical screening visit, e.g., systolic blood pressure exceeding baseline reading by 20mmHg, diastolic blood pressure exceeding the baseline reading by 10mmHg, BP > 160/100, or resting pulse increased by 20 beats/minute from the baseline reading will be excluded from the study. Subjective side effects will be measured for 21 potential side effects (e.g., headache, nausea, nervousness, etc.) by having subjects rate the intensity of their symptoms using the following scale : 1 = none, 2 = mild, 3 = moderate, 4 = severe. A qualified registered nurse is present throughout the entire session. Furthermore, thorough emergency plans have been implemented in conjunction with the Children's Hospital of Eastern Ontario (e.g. code blue) and the University of Ottawa should a crisis arise. In addition, the research unit has been equipped with a complete first aid unit cart along with an automated external defibrillator in which all the employees have been trained to operate. All employees are also required to maintain a valid CPR-C.

Each participant will be supplied with a "study enrollment card" that will have the study title, along with the emergency contact information for the CHEO pharmacy technician (in control of study blinding) and for the Qualified Investigator (Principal Investigator-PI ). This card will act as a safeguard if the participant seeks emergency medical help where it is required to know whether they have been taking drug or placebo, thereby acting as an aid in the clinical judgment to stop the treatment. The enrollment card will also act to tract if/when a participant needs to be unblinded to the treatment.

Trial Management and Monitoring

Management

The Children's Hospital of Eastern Ontario Clinical Research Unit (CHEO-CRU) will be the coordinating center for this study and the University of Ottawa will the other testing site. The Principal Investigator and the study coordinator, along with CHEO pharmacy, will be responsible for the day-to-day operations of the trial. CHEO-CRU will provide the CHEO pharmacy with the randomization table and will resultantly be the only persons who are unblinded. The randomization will take place once the Initial Screening Visit is completed and it is determined that the participant is eligible to participate. Therefore, each participant will have an equal chance of being randomized to drug or placebo using a computer generated random number program by a member of the CRU before entering into the Baseline 1 test day.

Treatment discontinuation

In the event that the subject is withdrawn from the study due to an AE, the AE will be recorded and reported, and the subject will be followed and treated until the abnormal parameter or symptom has resolved or stabilized. It is up to the clinician and the Data & Safety Monitoring Board to determine that the AE is either resolved or that it has reached a stable state, after which no further follow-up is necessary. Support for this determination will be documented. The reason for withdrawal from the study will be recorded on the appropriate case report form (CRF). If a subject is removed from the study, we will continue the scheduled follow-up with the subject's permission. There will be no changes to the follow-up schedule, except no study treatment/intervention will be administered. If at any point a subject no longer wishes to participate in follow-up, or after the three month follow-up telephone call, participation in the study will be complete. If new evidence emerges in the literature to indicate that our study dosage is unsafe, the study will be discontinued and all further qualifying patients will be offered the more effective/safer treatment.

Data Safety and Monitoring Board

The Data and Safety Monitoring Board (DSMB) is an independent group of experts who will function independently and at arm's length from the Study Investigators and the Steering Committee of the Study. The primary responsibilities of the DSMB are as follows:

1. Review and evaluate the accumulated study data for participant safety
2. Make recommendations to the Steering Committee based on these reviews regarding the continuation, modification or termination of the trial
3. DSMB members must maintain strict confidentiality concerning all privileged trial results, and during all phases of DSMB review and deliberations.
4. No member of the DSMB should have a direct involvement with the conduct of the study. No member should have financial, proprietary, professional or other interests that may affect impartial, independent decision-making by the DSMB.

   The DSMB will be notified of all serious unexpected adverse drug reactions and all deaths within 5 working days of knowledge of the SAE. It is the Qualified Investigator's responsibility to ensure that the DSMB is apprised of all new safety information relevant to the study.

   The DSMB will be scheduled on a regular basis and as often as necessary. Regular reviews will be conducted yearly and focused primarily on safety issues. A designated third party analysis (prepared by a study statistician) will be delivered to the DSMB two weeks prior to any scheduled review. Prior to study initiation, DSMB members will review study protocols, informed consents, Data and Safety Monitoring Plans and other relevant documents as needed (case report forms, manual of procedures, etc.). During the study, DSMB members will review all study protocol amendments.

   Adverse Events (AE's) and Serious Adverse Events (SAE's)

   Adverse Events

   Adverse events (AEs) are defined as any symptom, sign, illness or experience that occurs while participating in the study, including both during admission and as an outpatient. Abnormal clinical results will be considered to be adverse events if the abnormality:
   * results in study withdrawal
   * is associated with clinical signs or symptoms
   * leads to additional treatment or to further diagnostic tests
   * is considered by the investigator or Data & Safety Monitoring Board to be of clinical significance.

   Serious Adverse Event (SAE)

   A SAE is any adverse event that at any dose:
   * results in death
   * is life-threatening
   * requires inpatient hospitalization or prolongation of existing hospitalization
   * results in persistent or significant disability or incapacity
   * results in a congenital anomaly/birth defect
   * other serious (important event)
   * prolonged hospitalization, significantly beyond the expected length of stay
   * important medical events

   Serious Unexpected Adverse drug Reactions are SAEs that are likely to be related to the study drug.

   Medical and scientific judgment should be exercised in deciding whether expedited reporting is appropriate in other situations such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent one of the events listed above.

   Serious Adverse Event Reporting

   What to Report
   * Any SAE that meets the definition of a Reportable Serious Adverse Event
   * All life-threatening or fatal adverse events with an attribution of possible, probable, or definite

   The Sponsor Investigator will notify Health Canada (Office of Clinical Trials) for those events which meet regulatory requirements for expedited reporting, (i.e. events which are BOTH serious AND unexpected), AND which are thought to be related to protocol treatment (or for which a causal relationship with protocol treatment cannot be ruled out).

   Adverse Drug Reaction (ADR) report must be filed in the cases:
   * where the ADR is neither fatal nor life-threatening, within 15 days after becoming aware of the information
   * where it is fatal or life-threatening, immediately where possible and, in any event, within 7 days after becoming aware of the information
   * within 8 days after having informed Health Canada of the ADR, submit as complete as possible, a report which an assessment of the importance and implication of any findings

   This includes all serious events that are unexpected and related (i.e. possibly, probably, or definitely) to protocol therapy. Investigators must notify their Research Ethics Boards (REBs) and documents related to submission must be retained in the study binder on site.

   The submission of these events to the local ethics board should be done as soon as possible (within 30 days) or per local REB requirements. REB submissions greater than 90 days from the date of notification will be regarded as delinquent and a major deficiency will be assigned.

   Important medical events are those that may not be immediately life threatening, but are clearly of major clinical significance. They may jeopardize the subject, and may require intervention to prevent one of the other serious outcomes noted above.

   Monitoring of AE's/SAE's:

   Any AE that occurs between the time a study participant/parent signs the informed consent form and the time he/she completes the telephone follow-up (or at the time of early discontinuation of the subject from the study for any reason) will be captured and recorded. At each contact with the subject, the investigator (or designate) will seek information on adverse events by specific questioning and, as appropriate, by examination.

   The intensity of an AE is assessed as mild (usually transient in nature and generally not interfering with normal activities), moderate (sufficiently discomforting to interfere with normal activities), and severe (prevents normal activities).

   The maximum clinical intensity of all adverse events will be classified as:
   * Mild: Signs and symptoms that can easily be tolerated or ignored.
   * Moderate: Symptoms that cause discomfort but are tolerable; they cannot be ignored and affect concentration.
   * Severe: Symptoms that affect usual daily activity.

   The attribution of all adverse events will be classified as:
   * Unrelated to investigational agent/intervention

     * Not related The AE is clearly not related to the intervention
     * Doubtful The AE is not likely to be related to the intervention
   * Related to investigational agent/intervention

     * Possible The AE may be related to the intervention
     * Probable The AE is likely related to the intervention
     * Definite The AE is clearly related to the intervention

   An adverse drug reaction (ADR) is any untoward medical occurrence that the PI determines is likely related to the study drug (attribution of possible, probably, or definite).

   Feasibility

   There are no field studies looking at the effects of MPH on food intake (neither as a main outcome nor secondary outcome). Therefore, our only way of estimating effects sizes is extrapolating from our previous laboratory studies. In a laboratory study by the investigators, an effect size of .93 was attained in 9 obese adult males for the primary outcome of food intake with mean energy intake in kilocalories for MPH (0.5 mg/kg) and placebo of 843.5 + 393.4 and 1095.9 + 271.1, respectively. In a second study in 14 normal weight adult males and females, an effect size of .69 was attained, favouring MPH (0.5 mg/kg) for food intake in an ad libitum buffet meal with mean difference in kcals of -133 (1099 for MPH minus 1232 for placebo), with a standard deviation of 192.0 kcals for the paired differences based on t-tests. Based on the more conservative effect size of .69, it would be possible to detect a significant difference in kcals consumed over a 60-day period between MPH and placebo using a paired t-test with an alpha of 0.05, power of 0.80, with 18 participants per group. Thus, the plan to include 40 participants per group should enable the investigators to look at trends on other energy balance (secondary outcome) variables, accounting for an expected drop-out of 5-10%. The plan is to run 3 new participants/month, thus the experimental part of the study should last approximately 14 months.

   Role of Investigators/Staff

   Philippe Robaey, as Principal Investigator, is a physician and child Psychiatrist and Director of the ADHD clinic at CHEO. He has many years of clinical and research experience with MPH. Dr. Robaey will be responsible for the medical aspects of the study such as prescribing the study medication under double blind conditions, as well as overseeing the evaluation of vital sign and side effects of MPH. Dr. Eric Doucet, as Co-Principal Investigator (C0-PI) is a Full Professor of Human Kinetics at University of Ottawa, Faculty of Health Sciences. Dr. Doucet is an expert in the measurement of energy balance measures using the proposed methods. The study of the adult population will be conducted in Dr. Doucet's Behavioural Metabolic Research Unit, where our previous MPH cross-over trial was done, and he will oversee the coordination and supervision of the experimental testing procedures. Dr. Gary Goldfield, as Co-Principal Investigator (CO-PI), is a clinical psychologist and Investigator with the Healthy Active Living and Obesity Research Group at the CHEO Research Institute. He will oversee the assessment of psychiatric inclusion criteria evaluated by questionnaire and structured clinical interview, as well as the measurement of the reinforcing (rewarding) value of food. Dr. Jameason Cameron, as co-Principal investigator, is a postdoc and a research coordinator at CHEO. He has extensive experience with feeding studies and weight loss trials, and measures of food reward and smell function. Dr. Cameron will be responsible for the day-to-day testing and to supervise the PhD student who will be co-coordinating the study.

   Statistical Analysis

   Differences between groups (MPH vs. placebo) in energy intake and energy expenditure variables, as well as body weight, impulsivity, olfaction, hunger, satiety, and the reinforcing value of food will be evaluated by paired t-tests and repeated measures analyses of variance (ANOVA). Hypotheses of mechanisms linking MPH and reduced food intake and weight loss via reduced food reward will be explored using multiple regression mediational analyses as described by Baron and Kenny.

   Data Management

   All "source document" data collected from the study visits, except data that would indicate randomization assignment, will be maintained in a secure location within the Children's Hospital of Eastern Ontario. The investigator will verify that all data entries in the CRF are accurate and correct. Data collection is the responsibility of the research staff at the site under the supervision of the Principal Investigator. During the study the investigator will maintain complete and accurate documentation for the study and keep all original source documents. All adverse events will be graded, assessed by severity and causality and reviewed by the site investigator. Original subject records (source documents) will be reviewed during the course of the monitoring to verify the accuracy of the CRF's. This review will be conducted according to the peer monitoring plan. The Investigator(s) institutions(s) will permit trial-related monitoring, audits, REB(s) review and regulatory inspections(s) by providing direct access to source data and documentation. The medical (hospital/practice) records for each patient should contain information to provide a means by which study data can be verified. Patient information collected electronically will be available for review when the study site is monitored or audited. Entry of these data in SPSS will be performed primarily by the PhD student, but partly by the co-Principal investigators. Subjects will be assigned a code number to maintain blinding to data management staff, with the corresponding list of names associated with subject codes kept by the pharmacist in a secure filing cabinet. Databases will be stored on a secure server, with nightly backup.

   Publication Plan

   By the end of the second year of the study the investigators plan on publishing 2 peer-review articles, one at the international journal Physiology and Behavior highlighting the secondary metabolic outcomes, and the other at the American Journal of Clinical Nutrition, highlighting the main outcome of the influence of MPH on appetite.

   Ethical Considerations

   This study will be conducted according to Canadian and international standards of Good Clinical Practice and the Health Canada, Food and Drug Act, Part C, Division 5, Drugs for clinical Trials Involving Human Subjects, and in full conformance with principles of the "Declaration of Helsinki". The CHEO research institute policies and standard operating procedures will also be followed. This protocol and any amendments will be submitted to the CHEO REB for formal approval to conduct the study. The decision of the REB concerning the conduct of the study will be made in writing to the investigator. All participants for this study will be provided a consent form and assent form if applicable, describing this study and providing sufficient information for participants to make an informed decision about their participation in this study. The consent form will be submitted with the protocol for review and approval by the REB. The formal consent of a participant, using the REB-approved consent form, will be obtained before that participant is submitted to any study procedure. The consent form must be signed by the participant or legally acceptable surrogate, and the investigator-designated research professional obtaining the consent.

ELIGIBILITY:
Inclusion Criteria:

* males and females 16 to 40 years old
* BMI in the obese category (above 29.9kg/m2)
* willing to comply with procedures, and sign informed consent forms
* able to swallow a placebo pill that will be used in the study (same size as study drug)

Exclusion Criteria:

* smoker (the main outcome is energy intake and smoking is known to impact appetite)
* known serious food allergies, including lactose
* history of previous MPH use or allergy to MPH
* history of ADHD or current diagnosis of an axis 1 psychiatric disorder (e.g., depression, panic disorder, schizophrenia) as measured by self-report, the Wender-Utah Rating Scale52-54 and the Beck Depression Inventory
* current use of antidepressants, thyroid medication, or any medication that could affect appetite
* high blood pressure
* pre-existing cardiovascular disorders including uncontrolled hypertension, angina pectoris, arterial occlusive disease, heart failure, cardiomypathies, myocardial infarction, and cardiac arrhythmia
* diabetes
* excessive use of alcohol or alcoholism, or current addictions to opiates, cocaine or stimulants as measured by the Drug Abuse Screening Test;
* not a restrained eater based on cut-score (11 or higher) on Three Factor Eating Questionnaire56
* glaucoma
* personal or family history of seizure disorders
* currently taking MAO inhibitors, pressor agents, coumarin, anticonvulsants, phenylbutazone, or tricyclic antidepressants
* history of thyroid disease
* personal or family history of motor tics or Tourettes's Syndrome
* not pregnant, as determined by commercially available pregnancy test taken by female participants prior to test dose of MPH.
* after the test dose of MPH, systolic blood pressure exceeding baseline reading by 20mmHg, diastolic blood pressure exceeding the baseline reading by 10mmHg, BP > 160/100, or resting pulse increased by 20 beats/minute from the baseline.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in Energy Intake | Measured three times over the course of 2 months (twice at baseline: once with and without study drug & once at final visit).
  Participant will be offered a lunch buffet that includes items they indicate are preferred. They will be able to eat as much or as little as they choose.

SECONDARY OUTCOMES:
Change in Energy Expenditure | Measured three times over the course of 2 months (twice at baseline: once with and without study drug & once at final visit).
  Indirect calorimetry measure: participant lies supine on a bed while a neoprene mask is attached to their face. Expired breath is captured by the metabolic cart to assess resting energy expenditure and the thermic effect of feeding.
Change in Body Weight | Measured two times over the course of 2 months (once at baseline & once at final visit).
  Participant stands on a weight scale.
Height | Measured at baseline.
  Participant stands next to a stadiometer; height will be used to determine BMI at baseline.
Height | Measured at final visit; height will be used to determine BMI at the final visit.
  Participant stands next to a stadiometer
Change in Body Mass Index | Measured two times over the course of 2 months (once at baseline & once at final visit).
  This measure is a conglomerate of body weight (kg) divided by height (meters squared)
Change in Impulsivity towards food and non-food reward as measured by reaction time on a computer task. | Measured three times over the course of 2 months (twice at baseline: once with and without study drug & once at final visit).
  A "go/no-go"computer task that measures reaction time to food and non-food cues with simple button-presses on a keyboard.
Change in Odour Detection Threshold measured with Sniffin' Sticks Odourized Pens | Measured three times over the course of 2 months (twice at baseline: once with and without study drug & once at final visit).
  Odourized pens, called Sniffin Sticks, are used to measure odour detection threshold for a non-toxic odourant called n-butanol.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Doucet, PhD, Study Chair — University of Ottawa; Philippe Robaey, MD, FRCPC, Principal Investigator — Childrens Hospital of Eastern Ontario-Research Inst
Locations (2):
- Canada (2):
  - Children's Hospital Of Eastern Ontario Research Institute, Ottawa, Ontario
  - University of Ottawa, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: Undecided
We have not made a plan to make IPD available. We do plan on publishing the findings, but as per normal scientific reporting, with deidentified data.